CLINICAL TRIAL: NCT03523273
Title: Pilot Study of the Effect of Liraglutide 3.0 mg on Weight Loss and Gastric Functions in Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Camilleri, MD (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Michael Camilleri, MD, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 15-001783 Part B; R56DK067071 (NIH); UL1TR000135 (NIH)
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Results first posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liraglutide (Experimental): Liraglutide initiated at 0.6mg S.C. daily for 1 week; subjects will return to the Clinical Research Unit (CRU) each week until an increase by 0.6 mg/day in weekly intervals to a dose of 3.0 mg/day is achieved. Once maintenance dose of 3.0 mg is achieved, subjects will return approximately every 4 weeks to obtain new supply of study medication.
  Interventions: Drug: Liraglutide
- Placebo (Experimental): Placebo initiated at 0.6mg S.C. daily for 1 week; subjects will return to the Clinical Research Unit (CRU) each week until an increase by 0.6 mg/day in weekly intervals to a dose of 3.0 mg/day is achieved. Once maintenance dose of 3.0 mg is achieved, subjects will return approximately every 4 weeks to obtain new supply of study medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — Initiate at 0.6mg S.C. daily for 1 week; subjects will return to the Clinical Research Unit (CRU) each week until an increase by 0.6mg/day in weekly intervals to a dose of 3.0 mg/day is achieved (~4 weeks). Once maintenance dose of 3.0 mg is achieved, subjects will return approximately every 4 weeks to obtain new supply of study medication.
  Other Names: Saxenda; Victoza
  Arms: Liraglutide
Drug: Placebo — Placebo administration will match the study drug.
  Arms: Placebo

SUMMARY:
This study is being done to assess the stomach emptying effect of a maximum dose of 3 mg Liraglutide compared to placebo in subjects who are overweight or obese. Liraglutide is a medication approved by the Food and Drug Administration (FDA) for routine clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese adults (≥30 kg/m^2 or ≥27 kg/m^2 with an obesity-related co-morbidity).
* Subjects residing within 125 miles of Mayo Clinic in Rochester, Minnesota.
* Healthy individuals with no unstable psychiatric disease and not currently on treatment for cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, or endocrine (other than hyperglycemia type 2 diabetes mellitus on metformin) disorders.
* The investigators plan to recruit equal proportions of men and women.
* Women of childbearing potential will be using an effective form of contraception, and have negative pregnancy tests within 48 hours of enrollment and before each radiation exposure. In addition, since liraglutide 3.0 mg is classified as Pregnancy Category X, monthly urine pregnancy testing will be performed in any female participant with childbearing potential.
* Subjects must have the ability to provide informed consent before any trial-related activities.

Exclusion Criteria:

* Weight exceeding 137 kilograms (safety limit of camera for measuring gastric volumes).
* Abdominal surgery other than appendectomy, cholecystectomy, Caesarian section or tubal ligation.
* Positive history of chronic gastrointestinal diseases, systemic disease that could affect gastrointestinal motility, or use of medications that may alter gastrointestinal motility, appetite or absorption, e.g., orlistat.
* Patients with a personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia-type 2.
* Patients with a past or current history of pancreatitis, gallstones, history of alcoholism, blood triglyceride levels >500 mg/dL.
* Significant untreated psychiatric dysfunction based upon screening with the Hospital Anxiety and Depression Inventory (HAD), a self-administered alcoholism screening test (AUDIT-C), and the Questionnaire on Eating and Weight Patterns (binge eating disorders and bulimia). If such a dysfunction is identified by a HAD score >11 on either the Anxiety or Depression subscales, or difficulties with substance or eating disorders, the participant will be excluded and given a referral letter to his/her primary care doctor for further appraisal and follow-up.
* Intake of any medication (except multivitamins), within 7 days of the study. Exceptions are birth control pill, estrogen replacement therapy, thyroxin replacement therapy and any medication administered for co-morbidities as long as they do not alter gastrointestinal motility including gastric emptying (GE) and gastric accommodation. For example, statins for hyperlipidemia, diuretics, β-adrenergic blockers, Angiotensin Converting Enzyme (ACE) inhibitors and angiotensin antagonists for hypertension, and metformin for type 2 diabetes mellitus or prediabetes are permissible. In contrast, resin sequestrants for hyperlipidemia (which may reduce GE and reduce appetite, α2-adrenergic agonists for hypertension, or other glucagon-like peptide-1 receptor agonists (GLP-1) receptor agonists (exenatide) or amylin analogs (pramlintide) are not permissible because they significantly affect GE and/or gastric accommodation.
* Delayed gastric emptying at 2 and 4 hours
* Hypersensitivity to the study medication, liraglutide
* Participate in highly intense physical activity program that could potentially interfere with study interpretation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liraglutide | Placebo
Started | 67 | 69
Completed | 59 | 65
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Placebo | Total
Number analyzed (Participants) | 67 | 69 | 136
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42 [32 to 51] | 37.2 [29.3 to 45.2] | 37.7 [30.8 to 49.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 59 | 118
  Male | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 60 | 65 | 125
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 67 | 69 | 136

OUTCOME MEASURES:

1. Primary Outcome: Gastric Emptying of Solids (T1/2)
Description: The time for half of the ingested solids to leave the stomach. Following a meal consisting of two eggs labeled with technetium Tc 99m sulfur colloid (1 mCi), gastric emptying of solids was assessed with scintigraphy imaging.
Time Frame: 5 weeks
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 67 | 69
minutes | 191.6 [137.0 to 241.0] | 105.9 [92.6 to 127.8]

2. Primary Outcome: Gastric Emptying of Solids (T1/2)
Description: as for outcome 1
Time Frame: 16 weeks
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 67 | 69
minutes | 154.4 [120.4 to 178.3] | 111.4 [97.3 to 132.9]

3. Secondary Outcome: Change in Weight at 5 Weeks
Description: Change in subject's weight, in kilograms
Time Frame: baseline, 5 weeks
Measure: Median (Inter-Quartile Range); unit: kilograms
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 67 | 69
kilograms | -3.8 [-4.8 to -2.5] | 0.1 [-1.5 to 1.4]
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Weight at 16 Weeks
Description: Change in subject's weight, in kilograms
Time Frame: baseline, 16 weeks
Measure: Median (Inter-Quartile Range); unit: kilograms
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 67 | 69
kilograms | -5.8 [-8.3 to -3.9] | 0.0 [-3.1 to 2.1]
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority; p = 0.033, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Satiety
Description: Subjects self-reported fullness after eating as much of a prescribed meal measured by kilocalories of food consumed.
Time Frame: 16 weeks
Measure: Median (Inter-Quartile Range); unit: kilocalories
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 67 | 69
kilocalories | 647.5 [472.4 to 826.4] | 793.7 [624.6 to 1019.3]

6. Secondary Outcome: Satiation Volume to Fullness
Description: Subjects ingest Ensure 300mL drink meal at a constant rate of 30mL/min until self-reported fullness and volume consumed will be measured in milliliters (mL).
Time Frame: 16 weeks
Measure: Median (Inter-Quartile Range); unit: milliliters (mL)
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 67 | 69
milliliters (mL) | 622.1 [496.7 to 746.6] | 746.6 [497.7 to 871.0]

7. Secondary Outcome: Maximum Satiation
Description: Subjects ingest Ensure 300mL drink meal at a constant rate of 30mL/min until they reach maximum or unbearable fullness. Volume consumed will be measured in milliliters (mL).
Time Frame: 16 weeks
Measure: Median (Inter-Quartile Range); unit: milliliters (mL)
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 67 | 69
milliliters (mL) | 974.4 [746.6 to 1156.3] | 1119.8 [995.4 to 1430.9]

8. Secondary Outcome: Fasting Gastric Volume Prior to Meal
Description: Gastric fasting volume was measured prior to a meal of 300 mL Ensure drink using noninvasive single photon emission-computed tomography (SPECT) of the stomach.
Time Frame: 16 weeks
Measure: Median (Inter-Quartile Range); unit: milliliters (mL)
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 67 | 69
milliliters (mL) | 221.2 [187.7 to 269.8] | 191.5 [176.5 to 231.5]

9. Secondary Outcome: Gastric Volume After Meal
Description: Gastric volume was measured after a meal of 300 mL Ensure drink using noninvasive single photon emission-computed tomography (SPECT) of the stomach.
Time Frame: 16 weeks
Measure: Median (Inter-Quartile Range); unit: milliliters (mL)
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 67 | 69
milliliters (mL) | 629.1 [538.9 to 705.1] | 583.8 [549.8 to 667.7]

10. Secondary Outcome: Gastric Accommodation
Description: Measured in milliliters (mL), using the difference between the fasting gastric volume prior to the meal and the gastric volume after the meal.
Time Frame: 16 weeks
Measure: Median (Inter-Quartile Range); unit: milliliters (mL)
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 67 | 69
milliliters (mL) | 385.4 [332.6 to 445.2] | 391.8 [348.6 to 433.5]

ADVERSE EVENTS:
Time Frame: Adverse events will be collected from baseline to end of study participation for a total of approximately 18 weeks on all participants.
Arm/Group | Liraglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/69
Serious Adverse Events (participants affected / at risk) | 1/67 | 1/69
Other Adverse Events (participants affected / at risk) | 67/67 | 56/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=67) | Placebo (N=69)
Cholecystectomy for acute cholecystitis associated with gallstones (Gastrointestinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=67) | Placebo (N=69)
Nausea (Gastrointestinal disorders) | 40 (40) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 23 (23) | 6 (6)
Abdominal pain/discomfort (Gastrointestinal disorders) | 19 (19) | 4 (4)
Constipation (Gastrointestinal disorders) | 18 (18) | 4 (4)
Headache (General disorders) | 18 (18) | 10 (10)
Bruising at injection site (General disorders) | 13 (13) | 9 (9)
Bloating (General disorders) | 11 (11) | 5 (5)
Burping/Belching (General disorders) | 6 (6) | 0 (0)
Abdominal cramping (Gastrointestinal disorders) | 6 (6) | 3 (3)
Lightheaded (General disorders) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT03523273/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT03523273/ICF_001.pdf